CLINICAL TRIAL: NCT00307723
Title: A Tolerability and Efficacy Study of the Angiogenesis Inhibitor Bevacizumab in Combination With 5-Fluorouracil, Oxaliplatin, and External Beam Radiation Therapy Followed by Gemcitabine and Bevacizumab for Locally Advanced Pancreatic Cancer
Brief Title: Study of Bevacizumab in Combination With 5-FU, Oxaliplatin and External Beam Radiation Followed by Gemcitabine and Bevacizumab for Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Lawrence Blaszkowsky< MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 05-233
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: EBRT; advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Fluorouracil; Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen Level 1 (Experimental): Radiation/Oxaliplatin/5-FU
  Interventions: Drug: bevacizumab; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: gemcitabine; Procedure: External Beam Radiation Therapy
- Regimen Level 2 (Experimental): Radiation/Oxaliplatin/Bevacizumab/5-FU
  Interventions: Drug: bevacizumab; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: gemcitabine; Procedure: External Beam Radiation Therapy

INTERVENTIONS:
Drug: bevacizumab — Intravenously on days 1, 15 and 29 of the first cycle. Intravenously on days 1, 15 of each 28-day cycles for cycles 2-5.
Drug: 5-Fluorouracil — Continuous infusion on days 1-5, 8-12, 15-19, 22-26, 29-33 and 36-38 of cycle one.
Drug: Oxaliplatin — Intravenously on dasy 1, 8, 15, 22, 29, 36 of cycle one.
Drug: gemcitabine — Intravenously on days 1, 8, 25 of every 28-day cycle for cycles 2-5.
Procedure: External Beam Radiation Therapy — Monday through Friday ending on day 38 of cycle 1

SUMMARY:
The purpose of this study is determine the safety of bevacizumab, oxaliplatin, 5-FU, and gemcitabine in combination with external beam radiation therapy(Phase I portion) as well as to begin to collect information about whether this combination treatment is effective in treating patients with locally advanced pancreatic cancer (Phase II portion).

DETAILED DESCRIPTION:
* The combination of all three drugs and radiation treatment has never been given to people before, therefore, we are going to add just one additional drug at a time for safety reasons.
* The first group of participants (3-4) who enroll on the study will receive 5-FU, radiation therapy with the added drug oxaliplatin, this is called Regimen level 1. If these participants have few or easily manageable side effects, then another group of participants will be enrolled and will receive 5-FU, radiation, oxaliplatin with the addition of bevacizumab this is called Regimen level 2.
* The combination of study drugs and radiation will last about 6 weeks, this 6 week period is called a cycle 1.
* Regimen Level 1 will receive the following: oxaliplatin intravenously on days 1, 8, 15, 22, 29, and 36; 5-FU infused by a continuous infusion on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38; radiation therapy Monday-Friday to complete on day 38.
* Regimen Level 2 will receive the following; bevacizumab intravenously on days 1, 15, and 29; oxaliplatin intravenously on days 1, 8, 15, 22, 29 and 36; 5-FU infused by continuous infusion days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38; radiation therapy Monday-Friday to complete on day day 38.
* The following are tests and procedures that will be performed during cycle 1: physical examination; blood work, urine sample. perfusion CT scan on day 12 (for those participants enrolled at Massachusetts General Hospital).
* At the end of cycle 1, CT scans will be performed to evaluate the participants disease status before they receive combination gemcitabine and bevacizumab. If the scans show the tumor has reduced in size and can be surgically removed, then surgery will be scheduled and the patient will receive gemcitabine and bevacizumab about 4 weeks after the surgery. If the scans show the tumor can not be removed, the patient will receive the gemcitabine/bevacizumab combination about 4 weeks after completing cycle 1.
* Cycles 2-5 consist of: gemcitabine given intravenously on days 1, 8, and 15 every 28 days; bevacizumab given intravenously on days 1 and 15 every 28 days. During cycles 2-5 the following tests and procedures will be performed: physical examination including vital signs on day 1 and 15 of each cycle; blood work on days 1, 8 and 15 of each cycle; a urine sample on day 1 of each cycle; CT scans will be done every 2 cycles.
* It will take about 7 months to complete the study treatment (longer for those who have surgery after Cycle 1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically and radiologically confirmed locally advanced pancreatic ductal adenocarcinoma and have not received prior therapy
* Disease is measurable by CT scan
* Age >= to 18 years
* Life expectancy of 4 months or longer
* ANC >/= 1,500mm/cm3
* Hemoglobin >/= 9g/dl
* Platelet count >/= 100,000/cm3
* Total bilirubin </= 2 times control
* SGOT/SGPT </= 2.5 times upper limit of normal
* Serum creatinine < 2mg/dl
* No evidence of metastatic disease by laparoscopy

Exclusion Criteria:

* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk for complications
* No secondary malignancies other than non-melanoma skin cancers or carcinoma in-situ of the cervix within past 5 years
* Patients with pre-existing peripheral neuropathy of grade 2 or greater
* Pregnant or lactating women
* Current, recent (within 4 weeks of study entry) or planned participation in an experimental drug study
* Blood pressure of >150/100 mmHg
* Unstable angina
* New York Heart Association Grade II or greater congestive heart failure
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy,m or significant traumatic injury within 28 days prior to day 0
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0
* Urine protein creatinine ratio > or = to 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 0
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of the combination of bevacizumab, 5-FU, oxaliplatin, and EBRT for locally advanced pancreatic cancer | 2 years
to determine the survival of patients treated with this regimen.

SECONDARY OUTCOMES:
To determine the progression free survival
to determine the rate of conversion to resectability after treatment | 2 years
to asses the duration of response and response rate of this combination and
to evaluate the toxicities. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S. Blaszkowsky, MD, Principal Investigator — Massachusetts General Hospital